CLINICAL TRIAL: NCT05926648
Title: Form, Fit, and Function of INVSENSOR00061
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP-1077
Record Dates: First submitted 2023-05-30; First posted 2023-07-03 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Test Subjects (Experimental): All subjects who are enrolled into the test group and participate in data collection receive the noninvasive INVENSOR00061
  Interventions: Device: INVSENSOR00061

INTERVENTIONS:
Device: INVSENSOR00061 — Noninvasive pulse oximetry and pulse rate device

SUMMARY:
The objective of this study is to evaluate the form, fit, and function of INVSENSOR00061 when used on newborn and infant subjects 0-18 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a full-term newborn (37 weeks) - up to 18 months of age.
* The parent(s) or guardian(s) of minor subjects are able to read and communicate in English and understand the study and the risks involved.

Exclusion Criteria:

* Subject has underdeveloped skin.
* Subject has a skin condition and/or deformity at the planned application site, which would preclude sensor placement and measurements.
* Subject has an absence or deformities of limbs or severe edema, which would interfere with sensor application or prevent the proper fit of the sensors.
* Subject has any medical condition which in the judgment of the investigator and/or study staff, renders them ineligible for participation in this study or subject is deemed ineligible by the discretion of the investigator/study staff.

Ages: 0 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Subjects: All subjects who are enrolled into the test group and receive the noninvasive INVENSOR00061
  INVSENSOR00061: Noninvasive pulse oximetry and pulse rate device
Period: Overall Study
Arm/Group | Test Subjects
Started | 53
Completed | 52
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Test Subjects: All subjects who are enrolled into the test group and received the noninvasive INVENSOR00061.
  INVSENSOR00061: Noninvasive pulse oximetry and pulse rate device
Arm/Group | Test Subjects
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 52
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 3
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: INVSENSOR00061 SpO2 Accuracy
Description: The SpO2 accuracy of INVSENSOR00061 was determined by calculating the accuracy root mean squared (Arms) difference between the measured values (SpO2i) to the reference values (SpO2ref_i) in accordance with ISO-80601-2-61.
  Arms= √(∑(i=1 to n) ((SpO2_i-SpO2ref_i )^2 ))/n
Time Frame: 2 hours
Population: 11 subjects not included in analysis due to incorrect sensor placement. 29 subjects not included in analysis due to absence of reference sensor used to calculate Arms.
Measure: Number; unit: % of SpO2
Groups:
- Test Subjects: All subjects who are enrolled into the test group and received the noninvasive INVENSOR00061 and the reference sensor.
  INVSENSOR00061: Noninvasive pulse oximetry and pulse rate device
Arm/Group | Test Subjects
Number analyzed (Participants) | 12
% of SpO2 | 1.02

ADVERSE EVENTS:
Time Frame: 2 hours to 48 hours
Arm/Group | Test Subjects
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT05926648/Prot_SAP_000.pdf